CLINICAL TRIAL: NCT06707012
Title: Efficacy of Metformin as an Adjunct to Standard Antidepressant Therapy in Treating Depression Among Obese Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fazaia Ruth Pfau Medical College (Other)
Responsible Party: Principal Investigator, Sadia khan, Dr. Sadia Khan MBBS resident FCPS Pharmacology, Fazaia Ruth Pfau Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: frpmc.edu.pk@sadiakhan12345678; FMC, University (Other: AIR UNIVERSITY)
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Depression
Keywords: Depression; oxidative stress; antidepressants; obesity
MeSH Terms: conditions — Depression; Obesity | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Study Design This is a comparative clinical study with randomized groups. Participants will be allocated to either the metformin group or the placebo group in conjunction with standard antidepressant therapy. Randomization will be achieved using computer generated numbers in 1:1 ratio.
  Metformin Group: Starting dose of 500 mg metformin once daily, titrated up to 2000 mg/day based on tolerance along with standard treatment of depression according to Maudsley guidelines.
  Placebo Group: Identical placebo tablets, following the same titration schedule as the metformin group along with standard treatment of depression
  Setting:
  At psychiatric Out Patient Department of Fazaia Ruth Pfau Medical College and Hospital Karachi Pakistan
  Study Duration:
  18 months
Who Masked: Participant, Investigator
Masking Description: This will be double blind study in which participant and investigator who prescribe the drug will be blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): We will prescribe metformin with starting dose of 500 mg metformin once daily, titrated up to 2000 mg/day based on tolerance along with standard treatment of depression according to Maudsley guidelines.
  Interventions: Drug: Metformin Hydrochloride
- placebo group (Placebo Comparator): Identical placebo tablets, following the same titration schedule as the metformin group along with standard treatment of depression
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Participants will be divided in 2 groups
  1 group will receive metformin and 2nd group will receive placebo
  Other Names: GLUCOPHAGE

SUMMARY:
To evaluate the efficacy of metformin as an adjunct therapy in improving depressive symptoms and metabolic markers in newly diagnosed obese depressed patients on standard antidepressant therapy.

investigator will compare between Two groups

1. metformin group 2 placebo group Primary outcome measure will be the improvement in depressive symptoms, indicating by a reduction in Hamilton Depression Rating Scale (HAM-D) scores. Secondary outcome measures will include the assessment of oxidative stress markers, specifically by measuring the increase in enzymatic activity of superoxide dismutase, catalase, and glutathione peroxidase Investigators hypothesize that the addition of metformin to standard antidepressant treatment will result in a significant reduction in symptoms of depression among newly diagnosed obese individuals.

DETAILED DESCRIPTION:
This is a comparative clinical study with randomized groups. Participants will be allocated to either the metformin group or the placebo group in conjunction with standard antidepressant therapy. Randomization will be achieved using computer generated numbers in 1:1 ratio.

Metformin Group: Starting dose of 500 mg metformin once daily, titrated up to 2000 mg/day based on tolerance along with standard treatment of depression according to Maudsley guidelines.

Placebo Group: Identical placebo tablets, following the same titration schedule as the metformin group along with standard treatment of depression.

Study will take place at psychiatric Out Patient Department of Fazaia Ruth Pfau Medical College and Hospital Karachi Pakistan

Investigators will recruit participants from the psychiatric outpatient department of PAF Hospital diagnosed with depression according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition for at least 2 weeks and having obesity. depression is assessed with help of Hamilton Depression Scale (HAM-D). Participants whose score is above 8 and will meet the inclusion criteria will be added in study.

Informed consent:

Participants who meets the criteria will be asked for written informed consent form and explain in detail about the study

Base Line Data Collection After taking informed consent, detailed history, physical examination, HbA1c and serum creatinine will be measured. Participants whose HbA1c results is below 5.7% and creatinine clearance is above 30% will be selected in the study. Investigators will assess HbA1c, serum creatinine levels at every 12 weeks' interval. Serum levels of antioxidant enzymes (superoxide dismutase, catalase, glutathione peroxidase) will measured in participants by using biochemical assays at baseline and at the end of the study.

Follow up visits Participants will be followed up six times throughout the study duration. 1st follow up visit will occur at 4th week to evaluate the response to treatment by using Hamilton depression rating scale for depression, as according to Maudsley guidelines initial response to treatment should be assessed within 4 weeks. Next follow ups will take place at every 6th week till 36 weeks to assess improvement in depression and changes in BMI.

ELIGIBILITY:
Inclusion Criteria:

* • Age >18 to <45 years

  * Gender: Both genders (Male and Female)
  * BMI >25
  * Diagnosis: Newly diagnose cases of depression (mild to severe)
  * HBA1C: Less than 5.7% (non-diabetic range)

Exclusion Criteria:

* Existing diabetes

  * Acute illnesses like acute kidney injury, recent history of myocardial infarction, acute liver injury
  * Intellectual disabilities or inability to understand due to any reason
  * Presence of Psychiatric disorders other than depression
  * Chronic kidney disease (eGFR < 45 mL/min/1.73 m²).
  * Use of any psychotropic medication within the past 6 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Decrease scoring of Hamilton depression rating scale | 18 months
  Primary outcome measure will be the improvement in depressive symptoms, indicating by a change in Hamilton Depression Rating Scale (HAM-D) scores. Decrease in the score will be considered as indicator of improvement in depression.
  0-7: Normal (no depression) 8-13: Mild depression 14-18: Moderate depression 19-22: Severe depression 23 and above: Very severe depression Investigators will compare the change in both groups.

SECONDARY OUTCOMES:
elevation in oxidative enzymes level (superoxide dismutase,catalase,glutathione peroxidase | 18 months
  Secondary outcome measures will include the change in oxidative stress markers, specifically by measuring the enzymatic activity of superoxide dismutase, catalase, and glutathione peroxidase. Increase in levels of enzymes will be considered as indicator of improvement of depression.
  investigators will compare the change in both groups.

OTHER OUTCOMES:
change in Basal Metabolic Rate | 18 months
  weight in kilograms and height in meters of the participants will be assessed at each follow up visit to identify change in basal metabolic rate and will compare between groups

CONTACTS AND LOCATIONS:
Overall Officials: sadia khan, MBBS, Principal Investigator — Fazaia Ruth Pfau Medical College
Locations (2):
- Pakistan (2):
  - Fazaia Rurh Pfau Medical College, Karachi, Sindh
  - Fazaia Ruth Pfau Medical College, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No
It will be shared if required by authority

REFERENCES:
- [Background] Guo M, Mi J, Jiang QM, Xu JM, Tang YY, Tian G, Wang B. Metformin may produce antidepressant effects through improvement of cognitive function among depressed patients with diabetes mellitus. Clin Exp Pharmacol Physiol. 2014 Sep;41(9):650-6. doi: 10.1111/1440-1681.12265. PMID 24862430
- [Background] Farooq S, Khan T, Zaheer S, Shafique K. Prevalence of anxiety and depressive symptoms and their association with multimorbidity and demographic factors: a community-based, cross-sectional survey in Karachi, Pakistan. BMJ Open. 2019 Nov 19;9(11):e029315. doi: 10.1136/bmjopen-2019-029315. PMID 31748286
- [Background] Heiskanen TH, Niskanen LK, Hintikka JJ, Koivumaa-Honkanen HT, Honkalampi KM, Haatainen KM, Viinamaki HT. Metabolic syndrome and depression: a cross-sectional analysis. J Clin Psychiatry. 2006 Sep;67(9):1422-7. doi: 10.4088/jcp.v67n0913. PMID 17017829
- [Background] Lang UE, Beglinger C, Schweinfurth N, Walter M, Borgwardt S. Nutritional aspects of depression. Cell Physiol Biochem. 2015;37(3):1029-43. doi: 10.1159/000430229. Epub 2015 Sep 25. PMID 26402520
- [Background] Luppino FS, de Wit LM, Bouvy PF, Stijnen T, Cuijpers P, Penninx BW, Zitman FG. Overweight, obesity, and depression: a systematic review and meta-analysis of longitudinal studies. Arch Gen Psychiatry. 2010 Mar;67(3):220-9. doi: 10.1001/archgenpsychiatry.2010.2. PMID 20194822
- [Background] Lee A, Morley JE. Metformin decreases food consumption and induces weight loss in subjects with obesity with type II non-insulin-dependent diabetes. Obes Res. 1998 Jan;6(1):47-53. doi: 10.1002/j.1550-8528.1998.tb00314.x. PMID 9526970
- [Background] Seifarth C, Schehler B, Schneider HJ. Effectiveness of metformin on weight loss in non-diabetic individuals with obesity. Exp Clin Endocrinol Diabetes. 2013 Jan;121(1):27-31. doi: 10.1055/s-0032-1327734. Epub 2012 Nov 12. PMID 23147210
- [Background] AlHussain F, AlRuthia Y, Al-Mandeel H, Bellahwal A, Alharbi F, Almogbel Y, Awwad O, Dala'een R, Alharbi FA. Metformin Improves the Depression Symptoms of Women with Polycystic Ovary Syndrome in a Lifestyle Modification Program. Patient Prefer Adherence. 2020 Apr 15;14:737-746. doi: 10.2147/PPA.S244273. eCollection 2020. PMID 32346286
- [Background] Calkin CV, Chengappa KNR, Cairns K, Cookey J, Gannon J, Alda M, O'Donovan C, Reardon C, Sanches M, Ruzickova M. Treating Insulin Resistance With Metformin as a Strategy to Improve Clinical Outcomes in Treatment-Resistant Bipolar Depression (the TRIO-BD Study): A Randomized, Quadruple-Masked, Placebo-Controlled Clinical Trial. J Clin Psychiatry. 2022 Feb 1;83(2):21m14022. doi: 10.4088/JCP.21m14022. PMID 35120288
- [Background] Jitca G, Gall Z, Jitca CM, But MG, Majai E. Drug Repurposing of Metformin for the Treatment of Haloperidol-Related Behavior Disorders and Oxidative Stress: A Preliminary Study. Pharmaceutics. 2024 Mar 15;16(3):403. doi: 10.3390/pharmaceutics16030403. PMID 38543297